CLINICAL TRIAL: NCT04088097
Title: Development and Initial Efficacy Testing of a Cognitive-Behavioral Intervention to Treat Adolescent Binge Eating
Brief Title: Cognitive Behavioral Therapy for Adolescent Binge Eating and Loss of Control Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000024926; K23DK115893 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Binge Eating; Eating Disorders in Adolescence; Overweight and Obesity
Keywords: adolescent; cognitive-behavioral therapy; loss of control eating
MeSH Terms: conditions — Bulimia; Overweight; Obesity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Therapy (Experimental): Adapted Cognitive-Behavioral Therapy (CBT) for adolescents with binge eating or loss-of-control eating.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Adolescent Binge/Loss-of-Control Eating
- Control Condition (Other): Educational materials related to adolescent health and nutrition.
  Interventions: Other: Control Condition

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Adolescent Binge/Loss-of-Control Eating — Cognitive-behavioral therapy (CBT) developed for adolescents with binge eating or loss-of-control eating.
  Arms: Cognitive-Behavioral Therapy
Other: Control Condition — Educational and informational materials on adolescent health and nutrition.
  Arms: Control Condition

SUMMARY:
This study will develop and test a cognitive-behavioral intervention for adolescents with binge/loss-of-control eating.

DETAILED DESCRIPTION:
Youth who engage in binge eating or loss-of-control eating are at high risk for physical and mental health impairment, as well as excess weight gain. As there are few evidence-based treatments for adolescents with binge/loss-of-control eating, assessment and treatment have received minimal attention for adolescent patients. Among adults, cognitive-behavioral therapy (CBT) has a strong evidence base for binge-eating disorder. Adolescents have unique social, cognitive and emotional needs because of their developmental stage; unique treatment approaches are essential to meet these unique needs. This study will develop a new CBT treatment for adolescents with binge eating or loss-of-control eating (modifying adult CBT for binge-eating disorder, conducting interviews with adolescents about aspects of treatment that need to be modified, conducting an open series of patients who receive the active treatment). This study will also test the efficacy of the newly-developed CBT for adolescents with binge/loss-of-control eating versus a control group in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria: To be included, adolescents must:

1. Be in the age range ≥12 years old and ≤17 years old;
2. Have a BMI that places them above the 85th percentile based on their age and sex;
3. Report 2 episodes of binge/LOC eating (feeling a loss of control while eating) per month for the past 3 months;
4. Be otherwise-healthy youth (i.e., no uncontrolled or serious medical conditions);
5. Read, comprehend, and write English at a sufficient level to complete study-related materials;
6. Be available for participation in the study for 7 months.

Exclusion Criteria: Prospective participants will be excluded if the adolescent:

1. Has a medical or psychiatric condition that would require hospitalization or intensive care (e.g., neurological disorder, psychotic disorders, suicidality);
2. Has a medical or psychiatric condition that would prohibit them from engaging in behavioral treatment or moderate physical activity (e.g., cardiovascular problems);
3. Has uncontrolled medical condition(s) (e.g., uncontrolled diabetes or hypertension);
4. Is pregnant or breastfeeding;
5. Is taking medication(s) or participating in treatment(s) that could influence weight or appetite;
6. Began taking hormonal contraceptives less than 3 months prior;
7. Has a developmental or cognitive disorder (e.g., autism spectrum disorder);
8. Has a concurrent feeding/eating disorder (e.g., bulimia nervosa); or
9. Is participating in another clinical research study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy | Control Condition
Started | 25 | 25
Completed | 23 | 21
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy | Control Condition | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.20 (1.66) | 14.88 (1.33) | 14.54 (1.53)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 8 | 11 | 19
  Female | 17 | 13 | 30
  Non Binary | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 17 | 18 | 35
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
Binge Eating Episodes [Mean (Standard Deviation); unit: episodes of behavior] | 12.04 (9.19) | 13.57 (19.11) | 12.77 (14.62)

OUTCOME MEASURES:

1. Primary Outcome: Binge (Loss-of-control) Eating Episode Frequency
Description: Eating episodes will be assessed by questionnaire (Eating Disorder Examination questionnaire)
Time Frame: Post (4 months)
Measure: Mean (Standard Deviation); unit: episodes of behavior
Arm/Group | Cognitive-Behavioral Therapy | Control Condition
Number analyzed (Participants) | 21 | 19
episodes of behavior | 1.52 (2.09) | 6.05 (10.35)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy vs Control Condition; Test type: Superiority; p = .01, ANOVA

2. Primary Outcome: Weight (e.g., Percent Loss)
Description: Percent BMI change
Time Frame: Post (4 months)
Measure: Mean (Standard Deviation); unit: percentage of baseline BMI
Arm/Group | Cognitive-Behavioral Therapy | Control Condition
Number analyzed (Participants) | 21 | 20
percentage of baseline BMI | .02 (.13) | .01 (.06)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy vs Control Condition; Test type: Superiority; p = .75, ANOVA

3. Secondary Outcome: Binge (Loss-of-control) Eating Episode Frequency
Description: Eating episodes will be assessed by questionnaire (Eating Disorder Examination Questionnaire)
Time Frame: Short-Term Follow-Up (3 months after end of treatment)
Measure: Mean (Standard Deviation); unit: episodes of behavior
Arm/Group | Cognitive-Behavioral Therapy | Control Condition
Number analyzed (Participants) | 23 | 17
episodes of behavior | 2.04 (2.92) | 5.94 (9.59)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Therapy vs Control Condition; Test type: Superiority; p = .03, ANOVA

4. Secondary Outcome: Weight (e.g., Percent Loss)
Description: Percent BMI change
Time Frame: Short-Term Follow-Up (3 months after end of treatment)
Measure: Mean (Standard Deviation); unit: percentage of baseline BMI
Arm/Group | Cognitive-Behavioral Therapy | Control Condition
Number analyzed (Participants) | 23 | 18
percentage of baseline BMI | .02 (.14) | .01 (.06)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Cognitive-Behavioral Therapy | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT04088097/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04088097/ICF_000.pdf